CLINICAL TRIAL: NCT04086901
Title: Dose Escalated Adaptive RadioTherapy - a Randomised Phase II Study of Definitive Chemo-radiotherapy in Locally Advanced Esophageal Cancer
Brief Title: Dose Escalated Adaptive RadioTherapy in Definitive Chemo-radiotherapy for Esophageal Cancer
Acronym: DART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New data show no effect of dose escalation and also poor recruitment
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DART
Record Dates: First submitted 2019-08-22; First posted 2019-09-12 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Cancer
Keywords: Radiotherapy; Dose escalation; Definitive chemo-radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation Arm (Experimental): Chemo-radiotherapy with radiotherapy dose escalation based on Flour-Deoxy-Glucose /Positron Emissions Tomografi (FDG/PET) scans
  Interventions: Radiation: Radiotherapy dose escalation
- Standard (No Intervention): Standard chemo-radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy dose escalation — Flour-Deoxy-Glucose /Positron Emissions Tomografi (FDG-PET) scans will be used to identify and delineate the tumour sub-volumes with the highest tracer uptake to guide the dose-escalation. The dose to the Gross tumor volume (GTV) will be escalated to a high dose while clinical target volume (CTV) and planning target volume (PTV) will be treated with standard dose.
  Arms: Dose escalation Arm

SUMMARY:
In Denmark, 1000 new cases of esophageal and gastro-esophageal junction cancer occur every year. Surgery is the primary treatment for patients with localized disease who are considered medically and technically operable. For patients deemed non-resectable, definitive chemoradiotherapy is the treatment of choice, but despite treatment with curative intent, these patients have a poor prognosis, with a median survival of less than 20 months and a 5-year survival at 15-25% in clinical studies

This study will examine the effect of escalation of increasing the radiation dose to the most Positron Emissions Tomografi (PET) avid part of the tumour and lymph nodes compared to a standard uniform dose distribution.

DETAILED DESCRIPTION:
In Denmark, there are almost 900 new cases of oesphageal and gastro-esophageal junction (GEJ) cancer per year, with a 5-year survival rate below 20% for the entire group and a 5-year survival rate of approximately 40% for the curatively treated patients.

Surgery is the primary treatment for patients with localized disease who are considered medically and technically operable. For patients deemed non-resectable, definitive chemoradiotherapy is the treatment of choice, but despite treatment with curative intent, these patients have a poor prognosis, with a median survival of less than 20 months and a 5-year survival at 15-25% in clinical studies.

Survival is affected by several factors like stage, gender and comorbidity, but also by lack of local and regional tumour control. Several studies examined pattern of failure in patients with oesophageal cancer treated with definitive chemoradiotherapy. Most patients experience local failure, and most local failures were located in the Gross Tumor volume (GTV). These findings imply that future therapeutic strategies should focus on improving local control in order to increase successful treatment outcome, although care should be taken to ensure that this does not come at the cost of excess treatment related toxicity.

Strategies to overcome in-GTV failures include radiotherapy-sensitizing agents and dose escalation, the latter has been evaluated in several studies with heterogeneous results.

The role of Positron Emissions Tomografi/ComputerTomografi (PET/CT) in radiotherapy planning has been examined and the diagnostic value of PET/CT in oesophageal cancer is widely accepted, whereas the role in assessing tumour response to treatment is less well established. Flour-Deoxy-Glucose (FDG)-PET scans allow for measurement of changes in tumour cell metabolism that precede changes in tumour size, and reduction in FDG uptake during neoadjuvant therapy has been correlated with favourable outcomes in patients with oesophageal cancer.

PET-positive areas have been suggested as suitable targets for dose-escalation strategies, since studies suggested that high FDG uptake on pre-treatment PET/CT identifies tumour sub-volumes that are at greater risk of recurrence after chemoradiotherapy in patients with locally advanced oesophageal cancer.

The major concern in a dose escalation study is severe and potentially lethal normal tissue complications. Oesophageal cancer irradiation usually results in irradiation of the oesophagus, lungs and heart due to the anatomical tumour location, which may result in acute toxicities dominated by radiation pneumonitis and esophagitis (leading to inappropriate nutricial intake). Late toxicities include oesophageal fistula/ulcers, cardiac events, pulmonary fibrosis, or even deaths related to radiation exposure. Dose gradients between the target and normal tissue may be sharp, in order to limit the norml tissue dose and hence the risk of unacceptable toxicity, while maintaining high doses to the tumour.

Current study Previous studies have suggested that escalating the radiation dose to the GTV may provide improved local control, but requires great caution in relation to normal tissue irradiation to avoid unacceptable side effects. The investigators propose a study approach where both requirements will be met. FDG-PET scans will be used to identify and delineate the tumour sub-volumes with the highest tracer uptake to guide the dose-escalation. The dose to the GTV will be escalated to a high dose (63Gray (Gy) in the FDG-PET avid areas in the primary tumour and 60 Gy in the lymph nodes) while Clinical target volume (CTV) and Planning target volume (PTV) will be treated with standard dose. The patients will be randomized between this dose-escalated arm and a standard arm with 50Gy in 25 fractions. The total number of fractions will be 25 in both arms. Dose escalation will be limited by normal tissues constraints.

The study will be conducted with modern state-of-the-art radiotherapy techniques, including advanced dose calculation algorithms, daily image guidance, and adaptation of the treatment plan during treatment if needed. The participating centres must implement and comply with a quality assurance program in order to maintain high treatment quality in the study.

ELIGIBILITY:
Inclusion Criteria:

The patients must meet all of the following inclusion criteria to be included in the study:

* Patients with histologically verified squamous cell or adenocarcinoma (including signet cell carcinoma) of the oesophagus or GEJ.
* Multi-Disciplinary Team (MDT) assessment and treatment recommendation; deemed nonresectable and/or inoperable.
* TNM stage (8th edition): cT1-4a or cN+, cM0-1 (M1 disease limited to metastatic lymph nodes)
* Age ≥18 years.
* Performance status ≤2.
* Adequate cardiac, lung and renal function measured according to local guidelines.
* Adequate laboratory findings:

  * haematological: haemoglobin > 90 g/L, absolute neutrophil count (ANC) ≥ 1,5 x 109/L, platelets ≥ 75 x 109/L
  * hepatic: bilirubin ≤ 1.5 x ULN, ALAT ≤ 3 x ULN
  * renal: creatinine ≤ 1.5 x ULN
* Suitability to undergo curatively intended chemoradiation therapy.
* Ability to adhere to procedures for study and follow-up.
* Women must present a negative pregnancy test. Fertile men and women must use effective contraception. Fertile women included in the study must use oral contraceptives, intrauterine devices, depot injection of progestin subdermal implantation, a hormonal vaginal ring, or transdermal patch during the study treatment and one month after.
* Signed informed consent to participate in the study, including acceptance that dose plan and scans will be stored in a national dose plan bank, and the remaining data stored in a central database.
* A standard plan for radiotherapy with homogenous 50 Gy / 25 fractions, meeting all dose constraints for normal tissue, must be achievable.

Exclusion Criteria:

Patients who will meet one or more of the following exclusion criteria cannot be included in this study:

* Prior oncological treatment or surgical resection for the present disease
* Broncho-pulmonary fistula verified by bronchoscopy
* Any other active malignancies which may compromise study protocol or endpoints except for basal or squamous cell skin cancer
* Any unstable systemic disease (including clinically significant cardiovascular disease, unstable angina, New York Heart Association (NYHA) grade III-IV congestive heart, severe hepatic, renal or metabolic disease or active inflammatory bowel disease)
* Symptomatic peripheral neuropathy greater than grade 1 (CTCAE version 4.03)
* Any other serious or uncontrolled illness which in the opinion of the investigator makes it undesirable for the patient to enter the trial
* Severely decreased lung function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Loco-regional control | 12 months
  Loco-regional control evaluated with Flour-Deoxy-Glucose /Positron Emissions Tomografi (FDG-PET)

SECONDARY OUTCOMES:
Acute and late toxicity | 5 years
  Acute and late toxicity during and after treatment and at follow-up visits
Overall survival | 1 and 5 years
  Number of patients surviving
Progression-free survival | 1 and 5 years
  Survival without disease progression
Hospitalization | 12 months
  Time spent at hospital and number of hospitalizations due to radiation-induced toxicity
Mean and maximum dose distributions | 6 months
  Mean and maximum doses for all organs at risk will be compared between proton therapy (in silico) and (clinical) IMRT/VMAT photon therapy.
Dose distributions | 6 months
  V5, V10, V15, V20, V25, V30, V35, V40, V45 and V50 for all organs at risk will be compared between proton therapy (in silico) and (clinical) IMRT/VMAT photon therapy.
Pattern of failure in GTV-T | 5 years
  Number of Participants with failure in the Gross tumor volume-tumor (GTV-T)
Pattern of failure in GTV-N | 5 years
  Number of Participants with failure in the Gross tumor volume-nodes (GTV-N)
Pattern of failure in GTV-PET | 5 years
  Number of Participants with failure in Gross tumor volume-PET avid (GTV-PET)
Pattern of failure in CTV | 5 years
  Number of Participants with failure in the clinical target volume (CTV)
Pattern of failure in PTV | 5 years
  Number of Participants with failure in the Planning target volume (PTV)
Pattern of failure outside PTV | 5 years
  Number of Participants with failure in the outside the Planning target volume (PTV)
Stability of the FDG-PET signal, intensity | 12 months
  Changes in FDG-PET signal measured in terms of intensity
Stability of the FDG-PET signal, shape | 12 months
  Changes in FDG-PET signal measured in terms of shape
Stability of the FDG-PET signal, heterogeniety | 12 months
  Changes in FDG-PET signal measured in terms of heterogeniety
Correlation between loco-regional progression after treatment and changes in FDG-PET uptake pattern during standard and dose-escalated radiotherapy. | 12 months
  Response will be measured based on PERCIST and using radiomics characterizing the tumour in terms of uptake intensity, shape, and volumes.
Treatment completion rate | 12 months
  Number of patients completing all radiotherapy treatments and receiving at least one cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hanna R Mortensen, MD PhD, Principal Investigator — Aarhus University Hospital and Aarhus University
Locations (3):
- Denmark (3):
  - Rigshospitalet, Copenhagen, Capital Region
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Odense Universityhospital, Odense, Fyn

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Derived] Sakanaka K, Ishida Y, Fujii K, Ishihara Y, Nakamura M, Hiraoka M, Mizowaki T. Radiation Dose-escalated Chemoradiotherapy Using Simultaneous Integrated Boost Intensity-Modulated Radiotherapy for Locally Advanced Unresectable Thoracic Oesophageal Squamous Cell Carcinoma: A Single-institution Phase I Study. Clin Oncol (R Coll Radiol). 2021 Mar;33(3):191-201. doi: 10.1016/j.clon.2020.07.012. Epub 2020 Aug 4. PMID 32768158